CLINICAL TRIAL: NCT07025265
Title: The Effect of Antenatal Education Based on the Breastfeeding Self-Efficacy Theory and Postpartum Follow-Up Counseling on Breastfeeding Self-Efficacy and Attitudes in Adolescent Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hatice Nur Özgen, PhD Candidate in Obstetrics and Gynecology Nursing, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THESIS-2025-001
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Pregnancy; Breastfeeding; Self-Efficacy
Keywords: Adolescent Mothers; Breastfeeding Counseling; Prenatal Education; Postpartum Follow-Up; Lactation
MeSH Terms: conditions — Breast Feeding | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: This study follows a parallel interventional model where adolescent pregnant women are assigned to either the intervention group, receiving breastfeeding self-efficacy theory-based antenatal education and postpartum follow-up counseling, or the control group, receiving routine perinatal care. Outcomes related to breastfeeding self-efficacy and attitudes are compared between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Breastfeeding Self-Efficacy-Based Education and Counseling) (Experimental): Participants in this group will receive breastfeeding self-efficacy theory-based antenatal education and postpartum follow-up counseling. The education will be provided during the antenatal period, followed by weekly reminder and encouragement text messages until birth. Postpartum, participants will receive home visits in the first week for counseling and follow-up calls in the 2nd, 3rd, and 4th weeks.
  Interventions: Behavioral: Breastfeeding Self-Efficacy-Based Education and Counseling
- Control Group (Routine Perinatal Care) (No Intervention): Participants in this group will receive standard perinatal care without additional breastfeeding education or counseling. Postpartum data will be collected in the 4th week via a follow-up phone call.

INTERVENTIONS:
Behavioral: Breastfeeding Self-Efficacy-Based Education and Counseling — his intervention consists of breastfeeding self-efficacy theory-based education provided during the antenatal period. The education covers key factors affecting maternal breastfeeding self-efficacy, including previous experiences, vicarious learning, social support, and psychological responses. Weekly reminder and encouragement text messages will be sent until birth. Postpartum follow-up includes a home visit in the first week for counseling and phone-based follow-ups in the 2nd, 3rd, and 4th weeks.
  Arms: Intervention Group (Breastfeeding Self-Efficacy-Based Education and Counseling)

SUMMARY:
Adolescence is the period between the ages of 10 and 19, during which individuals undergo physiological, biological, psychological, and social development, transitioning from childhood to adulthood. Pregnancies occurring during this period are defined as adolescent pregnancies. In developing countries, approximately 21 million adolescent pregnancies occur annually among individuals aged 15-19, resulting in around 12 million births. According to national demographic data, a certain percentage of adolescent women have already started childbearing. Pregnancies occurring during this stage, when physical and psychosocial development is still incomplete, bring various medical and social challenges.

Adolescent pregnancies are associated with increased maternal and fetal mortality and morbidity risks and are classified as high-risk pregnancies. Therefore, adolescent mothers require close follow-up during both the antenatal and postpartum periods. However, studies indicate that adolescent mothers often fail to attend regular antenatal check-ups, receive inadequate education on breastfeeding, and consequently feel unprepared for motherhood. They tend to have low breastfeeding self-efficacy and develop negative attitudes toward breastfeeding. In the postpartum period, they also experience difficulties in initiating and maintaining breastfeeding.

Research highlights the need for education and counseling for adolescent mothers during the antenatal and postpartum periods. Providing education on breastfeeding is particularly important for improving maternal and infant health outcomes. Current approaches to breastfeeding counseling involve face-to-face training provided by healthcare professionals in medical institutions, as well as various alternative methods such as home visits, online/web-based education portals, theory-based training, text messages, emails, and phone consultations. In breastfeeding counseling, it is essential to not only provide education but also ensure continuous follow-up. Monitoring the process is expected to increase adolescent mothers' breastfeeding self-efficacy, foster positive attitudes toward breastfeeding, and extend the duration of breastfeeding.

This study aims to assess the effects of antenatal education based on the Breastfeeding Self-Efficacy Theory and postpartum follow-up counseling on adolescent mothers' breastfeeding attitudes and self-efficacy. By enhancing their breastfeeding self-efficacy and attitudes, this study is expected to contribute to resolving challenges related to early initiation and continuation of breastfeeding in the postpartum period.

DETAILED DESCRIPTION:
Study Population and Sample

Population:

The study population will consist of adolescent pregnant individuals registered at Family Health Centers in Şanlıurfa, Turkey.

Sample:

The sample size and power calculation were performed using the G*Power 3.1.9.4 program. The study sample size was determined using breastfeeding self-efficacy data from previous research, and the required number of participants was calculated as a total of 90, with at least 45 participants in each group. The Type I error rate was set at 0.05, and the effect size was determined as 0.6039, based on the means and standard deviations between groups. The power analysis result was 0.80.

Study Design

Randomization:

Block randomization will be used to assign participants to intervention and control groups. Complete randomization will be performed through https://www.randomizer.org. Two computer-generated randomization sequences will be applied in a one-to-one manner.

Intervention Group During the prenatal period, breastfeeding education based on the Breastfeeding Self-Efficacy Theory will be provided, and any questions from participants will be answered. According to the theory, a mother's breastfeeding self-efficacy is influenced by four key variables: previous breastfeeding experiences, observational learning from others, social support, and psychological state.

Following the education session, weekly reminder and motivational text messages related to breastfeeding will be sent until delivery.

In the first postpartum week, a home visit will be conducted for counseling, addressing any concerns, and collecting data.

During postpartum weeks 2, 3, and 4, participants will receive telephone counseling, and final data collection will occur in the 4th week.

Control Group Adolescent pregnant individuals who visit the Family Health Center will have their baseline data collected but will not receive any intervention.

They will continue to receive routine perinatal education. Final data will be collected via telephone in the 4th postpartum week. Data Collection Tools Personal Information Form Postpartum Mother Information Form I and II Breastfeeding Attitude Evaluation Scale Antenatal Breastfeeding Self-Efficacy Scale - Short Form Postpartum Breastfeeding Self-Efficacy Scale - Short Form Quality Assurance Measures Data Validation and Monitoring: Data entry will be controlled according to predefined rules, and inconsistencies will be corrected.

Source Data Verification: Participant data will be cross-checked with medical records and other reliable sources.

Standard Operating Procedures (SOPs): Standardized procedures will be established for patient registration, data collection, analysis, and adverse event reporting.

Ethical Considerations Ethical approval and institutional permissions were obtained from the Harran University Clinical Research Ethics Committee and the Şanlıurfa Provincial Health Directorate. The study will be conducted with pregnant individuals who voluntarily agree to participate. Written and verbal informed consent will be obtained from all participants, who will have the right to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent pregnant individuals (ages 14-19)
* Singleton pregnancy
* Gestational age of at least 28 weeks at enrollment
* Planning to breastfeed postpartum
* Willing to participate in antenatal education and postpartum follow-up counseling
* Able to provide informed consent

Exclusion Criteria:

* Multiple pregnancy (twins, triplets, etc.)
* Maternal or fetal conditions contraindicating breastfeeding (e.g., galactosemia)
* Severe maternal complications (e.g., preeclampsia with severe features, placenta previa with bleeding)
* History of previous breastfeeding difficulties or conditions affecting lactation (e.g., breast surgery)
* Psychiatric disorders that may interfere with participation
* Inability to complete follow-ups due to planned relocation or other reasons

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Breastfeeding Self-Efficacy Score | Baseline (before intervention), Postpartum Week 4
  The primary outcome will be assessed using the Postpartum Breastfeeding Self-Efficacy Scale-Short Form (PBSES-SF). This scale evaluates maternal confidence in breastfeeding, with higher scores indicating higher breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Exclusive Breastfeeding Rate at Postpartum Week 4 | Postpartum Week 4
  The percentage of mothers exclusively breastfeeding their infants at postpartum week 4 will be recorded.

OTHER OUTCOMES:
Maternal Satisfaction with Breastfeeding Support | Postpartum Week 4
  A questionnaire will assess maternal satisfaction with breastfeeding education and postpartum counseling received.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran Unıversity, Sanliurfa, Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be shared due to ethical considerations and confidentiality agreements. Data will only be accessible to authorized researchers involved in the study.